CLINICAL TRIAL: NCT03508141
Title: Fibrinogen Concentrate vs Cryoprecipitate in Traumatic Haemorrhage in Children: A Pilot Randomised Controlled Trial
Brief Title: Fibrinogen Early In Severe Trauma studY Junior
Acronym: FEISTY Jnr
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gold Coast Hospital and Health Service (Other Government)
Collaborators: Emergency Medicine Foundation (Other); National Blood Authority (Other); Australian Red Cross (Other)
Responsible Party: Principal Investigator, Dr James Winearls, BSc (Hons), MBBS, MRCP, FCICM, Dr James Winearls, Consultant Intensivist GCUH, Gold Coast Hospital and Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEISTY Jnr 1
Record Dates: First submitted 2018-03-23; First posted 2018-04-25 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Trauma; Hemorrhage; Coagulopathy; Pediatrics
Keywords: Fibrinogen Concentrate; Cryoprecipitate
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Hemostatic Disorders | interventions — Fibrinogen; cryoprecipitate coagulum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibrinogen Concentrate (Experimental): Fibrinogen Replacement using Fibrinogen Concentrate as per ROTEM (FIBTEM) FIBTEM A5 0mm = 60mg/kg FC FIBTEM A5 1-4mm = 50mg/kg FC FIBTEM A5 5-6mm = 40mg/kg FC FIBTEM A5 7-8mm = 30mg/kg FC FIBTEM A5 9-10mm = 20mg/kg FC
  Interventions: Drug: Fibrinogen Concentrate
- Cryoprecipitate (Active Comparator): Fibrinogen Replacement using Cryoprecipitate as per ROTEM (FIBTEM) FIBTEM A5 0mm = 6ml/kg Cryoprecipitate FIBTEM A5 1-4mm = 5ml/kg Cryoprecipitate FIBTEM A5 5-6mm = 4ml/kg Cryoprecipitate FIBTEM A5 7-8mm = 3ml/kg Cryoprecipitate FIBTEM A5 9-10mm = 2ml/kg Cryoprecipitate
  Interventions: Drug: Cryoprecipitate

INTERVENTIONS:
Drug: Fibrinogen Concentrate — Experimental
  Other Names: Riastap
  Arms: Fibrinogen Concentrate
Drug: Cryoprecipitate — Comparator
  Arms: Cryoprecipitate

SUMMARY:
1. Haemorrhage in severe trauma is a significant cause of mortality and is potentially the most preventable cause of death in paediatric trauma patients
2. Trauma Induced Coagulopathy (TIC) is a complex coagulopathy associated with severe trauma
3. Hypo/dysfibrinogenaemia plays an important role in TIC
4. Early replacement of fibrinogen may improve outcomes
5. Fibrinogen replacement is potentially inadequate in standard fixed ratio Major Haemorrhage Protocols (MHP) utilising Plasma and/or Cryoprecipitate
6. The majority of centres utilise cryoprecipitate for additional fibrinogen supplementation as part of a MHP
7. Cryoprecipitate administration is often delayed (between 60 - 120 minutes) in a fixed ratio MHP
8. It is clear early intervention in severe traumatic haemorrhage is associated with improved outcomes - CRASH 2 and PROPPR studies
9. Increasing interest in the use of Fibrinogen Concentrate (FC) in severe bleeding but not supported by high level evidence
10. Benefits of FC - viral inactivation, known dose, easily reconstituted, can be administered quickly in high dose and stored at room temperature in the trauma resuscitation bay

12. No previous studies comparing FC and Cryoprecipitate in bleeding paediatric trauma patients 13. Fibrinogen supplementation will be guided by an accepted ROTEM targeted treatment algorithm 14. Pilot, multi-centre randomised controlled trial comparing FC to Cryoprecipitate (current standard practise in fibrinogen supplementation) 15. Hypothesis: Fibrinogen replacement in severe traumatic haemorrhage can be achieved quicker with a more predictable dose response using Fibrinogen Concentrate compared to Cryoprecipitate 16. It is imperative that robust and clinically relevant trials are performed to investigate fibrinogen supplementation in paediatric trauma patients before widespread adoption makes performing such studies unfeasible

ELIGIBILITY:
Inclusion Criteria:

1. Child affected by trauma (3 months to 18 years)
2. Judged to have significant haemorrhage OR predicted to require significant transfusion by the treating clinician
3. Activation of Local MHP or transfusion of emergency red blood cells (Pre-hospital or at Trauma Centre)

Exclusion Criteria:

1. Injury judged incompatible with survival
2. Randomisation unable to occur within 6 hours of hospital admission
3. Pregnancy
4. Known personal or parental objection to blood products
5. Known coagulation disorder (i.e. haemophilia, von Willebrand disease)
6. Previous dedicated fibrinogen replacement this admission
7. Pre-Trauma Centre dedicated fibrinogen replacement
8. Participation in competing study

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to administration of fibrinogen replacement from time of identification of hypofibrinogenaemia requiring fibrinogen replacement | 3 Hours
  Time to fibrinogen replacement

SECONDARY OUTCOMES:
Transfusion Requirements | Up to 48 hours after Trauma Unit presentation
  In number of units of Packed Red Blood Cells, Plasma, FC, Cryoprecipitate, Platelets, Prothrombin Complex Concentrate at 4, 6, 24, 48hrs
Duration of bleeding episode or time until surgical control | It is anticipated that haemorrhage control will be achieved within 12 hours
  Duration bleeding episode
Intensive Care Unit LOS | 1 Year
  ICU LOS
Hospital LOS | 1 Year
  Hospital LOS
Adverse Events | 1 Year
  Transfusion related adverse events, Sepsis, Multiple Organ Failure, Acute Renal Failure, Symptomatic Thromboembolic Complications
All Cause Mortality | Up to 90 Days
  Mortality at 4, 6, 24 hours and up to 90 days
Functional Outcomes GOS-E Paediatrics | Up to 90 Days
  Functional Outcome Measures at 60 and 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Shane George, MBBS, Principal Investigator — Lady Cilento Children's Hospital
Locations (10):
- Australia (10):
  - Westmead Childrens Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Lady Cilento Children's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Mackay Base Hospital, Mackay, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] George S, Wake E, Jansen M, Roy J, Maconachie S, Paasilahti A, Wiseman G, Gibbons K, Winearls J; FEISTY Investigators. Fibrinogen Early In Severe paediatric Trauma studY (FEISTY junior): protocol for a randomised controlled trial. BMJ Open. 2022 May 4;12(5):e057780. doi: 10.1136/bmjopen-2021-057780. PMID 35508351